CLINICAL TRIAL: NCT04428723
Title: Mechanisms of Hypoglycemia in Patients Without Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00000095
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypoglycemia
Keywords: Microbiome; DNA; Hormones; Genetics
MeSH Terms: conditions — Hypoglycemia | interventions — Blood Specimen Collection; Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — Blood and fecal samples will be stored for up to 5 years for future analyses of additional blood proteins and metabolites and microbiome species which may contribute to hypoglycemia. DNA will be stored for additional expanded genotyping, depending on results of targeted resequencing. Fecal samples and /or cultures from them may be used for mouse transfer experiments in the future. All samples will be labeled only with the study identifier (ID) and acrostic unique to each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypoglycemia, no upper gastrointestinal (GI) surgery: Males or females with hypoglycemia with neuroglycopenia, but no history of upper GI surgery, diabetes or prediabetes
  Interventions: Other: Entry of demographic and medical history data into a deidentified database; Genetic: Blood sample for DNA analysis; Diagnostic Test: Stool sample for microbiome analysis; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Continuous glucose monitoring; Diagnostic Test: activity monitor
- Hypoglycemia, with history of upper GI surgery: Males or females with hypoglycemia with neuroglycopenia, with history of upper GI surgery
  Interventions: Other: Entry of demographic and medical history data into a deidentified database; Genetic: Blood sample for DNA analysis; Diagnostic Test: Stool sample for microbiome analysis; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Continuous glucose monitoring; Diagnostic Test: activity monitor
- Controls, without hypoglycemia or upper GI surgery: Males or females with no history of upper gastrointestinal surgery, hypoglycemia, or diabetes.
  Interventions: Other: Entry of demographic and medical history data into a deidentified database; Genetic: Blood sample for DNA analysis; Diagnostic Test: Stool sample for microbiome analysis; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Continuous glucose monitoring; Diagnostic Test: activity monitor

INTERVENTIONS:
Other: Entry of demographic and medical history data into a deidentified database — Entry into repository for analysis.
Genetic: Blood sample for DNA analysis — Targeted resequencing of DNA to identify variants associated with hypoglycemia, comparing participants with hypoglycemia (both surgical and non-surgical) and healthy controls.
Diagnostic Test: Stool sample for microbiome analysis — Participants will be asked to provide a fecal sample, collected at home, which will be analyzed to determine the types of bacteria present in the feces.
Diagnostic Test: Mixed meal tolerance test — For a subset of participants: After an overnight fast, participants will be given a standard liquid mixed meal; blood samples will be collected at baseline (fasting) and at defined time points after a meal for metabolic and hormonal analyses.
  Other Names: Meal Testing
Diagnostic Test: Continuous glucose monitoring — A CGM sensor (Dexcom G4 or other professional version available at onset of study) will be placed in blinded (masked) mode, and will be worn for 10 days. Data will be analyzed to determine patterns of glucose during both day and night intervals.
Diagnostic Test: activity monitor — The activity monitor (Fitbit Charge 2) will be worn by participants for 10 days, to assess activity, concurrent with CGM sensor wear.

SUMMARY:
The goal of this study is to identify physiologic and molecular mechanisms that underlie hypoglycemia in the absence of diabetes (or medications that can cause hypoglycemia) and to investigate potential genetic and microbiome differences which contribute to hypoglycemia. We will test the hypothesis that hypoglycemia in the absence of diabetes is linked to genetic variation or the microbiome, and identify whether additional medical history or diagnoses are enriched in the population of patients with hypoglycemia.

DETAILED DESCRIPTION:
Although there are several conditions which have been identified that cause, or contribute to hypoglycemia, diagnosis can be challenging, as the physiologic, and molecular mechanisms are incompletely understood. Additionally, treatment options are relatively limited, and often incompletely effective and/or not well tolerated. Investigating the causative factors and mechanisms of hypoglycemia is important therefore in improving our understanding in order to develop new and more effective approaches to treatment.

The current study aims to:

1. more fully characterize clinical history and demographics in patients with diverse forms of hypoglycemia by creating and analyzing a patient database;
2. for a subset of patients, characterize metabolic and hormonal responses to a standard meal;
3. analyze DNA variants in individuals with hypoglycemia;
4. analyze differences in the intestinal microbiome in individuals with hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. For hypoglycemia group without a history of bariatric surgery: Males or females diagnosed with hypoglycemia with prior episodes of neuroglycopenia.
2. For hypoglycemia group with history of upper gastrointestinal surgery: Males or females diagnosed with ongoing hypoglycemia with prior episodes of neuroglycopenia.
3. For non-surgical controls only: Males or females with no history of upper gastrointestinal surgery and no history of hypoglycemia or diabetes.
4. Age 18-70 years of age, inclusive, at screening.
5. Willingness to provide informed consent and attend one study visit, with option to attend a second visit with mixed meal test, and follow all study procedures

Exclusion Criteria:

1. Active treatment with any diabetes medications except for acarbose;
2. Known insulinoma, gastrinoma, or other neuroendocrine tumor;

Additional exclusion criteria for those participating in optional Visit 2 (meal testing):

1. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
2. Hepatic disease, including serum alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
3. Congestive heart failure, New York Hear Association (NYHA) class II, III or IV;
4. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use;
5. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia;
6. Concurrent administration of β-blocker therapy;
7. History of a cerebrovascular accident;
8. Seizure disorder (other than with suspect or documented hypoglycemia);
9. Active malignancy, except basal cell or squamous cell skin cancers;
10. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
11. Major surgical operation within 30 days prior to screening;
12. Hematocrit < 33% (women) or <36% (men);
13. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
14. Blood donation (1 pint of whole blood) within the past 2 months;
15. Active alcohol abuse or substance abuse;
16. Current administration of oral or parenteral corticosteroids;
17. Pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intrauterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
18. Use of an investigational drug within 30 days prior to screening.

There will be no involvement of special vulnerable populations such as fetuses, neonates, pregnant women, children, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups: (1) patients with hypoglycemia, but without a history of bariatric or other gastrointestinal surgery, recruited from the Joslin Hypoglycemia Clinic, (2) patients with hypoglycemia and history of upper gastrointestinal surgery, recruited from the Joslin Hypoglycemia Clinic,(3) controls without hypoglycemia or surgery, recruited by local advertisement or from family members of patients with hypoglycemia. We plan to enroll patients with hypoglycemia continuously over the next 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Entry of medical history data into a deidentified database. | March 2020 through March 2025
  Medical history data will be entered into RedCap for analysis.
Entry of physical exam data into a deidentified database. | March 2020 through March 2025
  Pertinent physical exam data will be entered into RedCap for analysis.
Entry of laboratory data into a deidentified database. | March 2020 through March 2025
  Laboratory data will be entered into RedCap for analysis.
Entry of demographic data into a deidentified database. | March 2020 through March 2025
  Demographic data will be entered into RedCap for analysis.
Analysis of participant demographics and medical history, comparing the 3 study groups. | March 2025
  Demographic and medical history data will be summarized in RedCap and compared between groups using ANOVA or chi-square testing, depending on the variable analyzed.
Targeted resequencing of DNA to identify variants associated with hypoglycemia, comparing patients with hypoglycemia (both surgical and non-surgical) and healthy controls. | March 2025
  Sequence variants identified during targeted resequencing will be summarized and prevalence will be compared between groups and with population databases. Depending on results of targeted resequencing, additional expanded genotyping may be performed.
Analysis of microbiome, comparing study groups. | March 2025
  Microbiome will be characterized by sequencing to obtain metagenomic data and pathway analysis; all data will be adjusted for multiple comparisons.
Analysis of glucose patterns during masked continuous glucose monitoring (CGM), including time in range, time in hypoglycemia, time in hyperglycemia, comparing the study groups. | March 2025
  For a subset of participants who consent to participate in optional Visit 2, CGM data will be analyzed to assess mean, median, peak, and nadir sensor glucose values, glycemic variability (GV), severity and length of hypoglycemia (% time glucose <70, <60, <54 mg/dL), and number and duration of severe hypoglycemia (sensor glucose <54, duration >15 minutes) will be quantified. Metrics will be assessed over 24 hours and during daytime (6 AM to midnight) and nighttime (midnight to 6 AM) independently.
Analysis of metabolic responses during mixed meal testing. | March 2025
  For a subset of participants who consent to participate in optional Visit 2, magnitude of hypoglycemia will be correlated with metabolite levels during meal testing. Metabolites will be measured at set time points after the start of the mixed meal. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in metabolic responses. Data will be checked to ensure variables conform to assumptions of the analysis. Sensitivity analysis will determine whether missing data are randomly associated with clinical or experimental phenotypes, and assess the impact of missing data on conclusions. The relationship between clinical and metabolic variables will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.
Analysis of hormonal responses during mixed meal testing. | March 2025
  For a subset of participants who consent to participate in optional Visit 2, magnitude of hypoglycemia will be correlated with hormone levels during meal testing. Counterregulatory hormones will be measured at set time points after the start of the mixed meal. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in counterregulatory hormone responses. Data will be checked to ensure variables conform to assumptions of the analysis. Sensitivity analysis will determine whether missing data are randomly associated with clinical or experimental phenotypes, and assess the impact of missing data on conclusions. The relationship between clinical and hormonal variables will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.

SECONDARY OUTCOMES:
Relationship between metabolic responses and magnitude of hypoglycemia as determined by CGM. | March 2025
  This is for a subset of participants (non-surgical hypoglycemia and controls) participating in optional Visit 2. Magnitude of hypoglycemia will be correlated with metabolite levels during meal testing.
Relationship between hormonal responses and magnitude of hypoglycemia as determined by CGM. | March 2025
  This is for a subset of participants (non-surgical hypoglycemia and controls) participating in optional Visit 2. Magnitude of hypoglycemia will be correlated with counterregulatory hormone levels during meal testing.
Relationship between metabolic responses and microbiome. | March 2025
  This is for a subset of participants (non-surgical hypoglycemia and controls) participating in optional Visit 2. Metagenomic data will be correlated with metabolic responses during meal testing.
Relationship between hormonal responses and microbiome. | March 2025
  This is for a subset of participants (non-surgical hypoglycemia and controls) participating in optional Visit 2. Metagenomic data will be correlated with counterregulatory hormone responses during meal testing.

OTHER OUTCOMES:
Safety outcome- hyperglycemia and hypoglycemia during the study | March 2025
  Participants will be closely monitored and glucose levels will be checked regularly at set time points during optional Visit 2. Symptoms of hypoglycemia will also be assessed at set time points during visits, and as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data may be shared with other researchers with permission of local institutional review boards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of study results.
Access Criteria: Data will be shared with academic investigators with approval of local institutional review boards.

REFERENCES:
- See also: recruitment website with contact information — http://www.joslin.org/research/clinical-research/clinical-trials/

DOCUMENTS (1):
  • Informed Consent Form (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04428723/ICF_000.pdf